CLINICAL TRIAL: NCT01727388
Title: Prospective Randomized Study Comparing the Results of Digital Rectal Examination in the Supine and Lateral Decubitus
Brief Title: Informativeness to Digital Rectal Examination
Acronym: RIFIONA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI11-PR-REGIMBEAU; 2011-AO1485-36 (Other: ID RCB)
Record Dates: First submitted 2012-10-22; First posted 2012-11-16 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Colon Cancer; Upper Rectum Cancer; Diverticulitis; Rectal Bleeding; Hernia
Keywords: rectal examination; colorectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Diverticulitis; Gastrointestinal Hemorrhage; Hernia; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lateral decubitus (Experimental): The digital rectal examination is performed in lateral decubitus i.e. curled up position . The patient in left lateral decubitus if the examiner is right handed and right lateral decubitus if the examiner is left handed.
  Interventions: Procedure: lateral decubitus
- supine decubitus (Active Comparator): The digital rectal examination is performed supine, spread legs, feet on the examination table. The examiner is in the patient's right side if he is right handed and in the patient's left side if he is left-handed.
  Interventions: Procedure: supine decubitus

INTERVENTIONS:
Procedure: lateral decubitus
  Arms: lateral decubitus
Procedure: supine decubitus
  Arms: supine decubitus

SUMMARY:
Digital rectal examination is an act clinically performed daily by physicians and surgeons. It remains the key diagnostic test and directs the therapeutic management of cancer of the lower and middle rectum. It can be done in two main positions: lateral decubitus, and supine.

However, no randomized study in colorectal surgery is not interested in evaluating the best position to perform a full rectal exam.

ELIGIBILITY:
Inclusion Criteria:

* colon or upper rectum cancer operated or not
* recurrent of colon or upper rectum cancer
* rectal bleeding
* hernia

Exclusion Criteria:

* woman
* paraplegic man
* bedridden patient
* current or previous pelvic radiotherapy
* History of prostatectomy
* emergency

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
realization of a full digital rectal examination | The consult could be done prior to the surgery or one month after the surgery
  Full digital rectal examination is defined by a rectal examination for investigating the superior pole of the prostate, to examine the entire circumference and the rectal sphincter.

SECONDARY OUTCOMES:
assessment of sphincter according to the DRESS score | The consult can be performed prior to the surgery or one month after the surgery
  This score assesses the sphincter tone at rest and during exercise. This score classes the sphincter tone in both situations: tone undetectable (score = 0) to hypertonic sphincter that does not allow the introduction of a finger (score = 5)
missing information during the rectal examination | The consult can be performed prior to the surgery or one month after the surgery
  This analysis aims to determine what information is missing most often in one group compared to another (height to digital rectal examination, circumference of the digital rectal examination , assessment of sphincter tone)
Conversion rate decided by the examiner | The consult can be performed prior to the surgery or one month after the surgery
  the conversion rate decided by the examiner corresponds to the switch from one position to another
Evaluation of the position by the patient | The consult can be performed prior to the surgery or one month after the surgery
  After the digital rectal examination, the examiner shows the patient a picture of the two positions and ask him the question: which position is the most embarrassing?

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Amiens Universitary Hospital, Amiens
  - Beauvais General Hospital, Beauvais

REFERENCES:
- [Result] Sabbagh C, Mauvais F, Vecten A, Ainseba N, Cosse C, Diouf M, Regimbeau JM. What is the best position for analyzing the lower and middle rectum and sphincter function in a digital rectal examination? a randomized, controlled study in men. Dig Liver Dis. 2014 Dec;46(12):1082-5. doi: 10.1016/j.dld.2014.08.045. Epub 2014 Sep 22. PMID 25245464